CLINICAL TRIAL: NCT04418531
Title: A Pilot Study to Explore the Efficacy and Safety of Rescue Therapy With Antibodies From Convalescent Patients Obtained With Double-filtration Plasmapheresis (DFPP) and Infused in Patients With Coronavirus Disease 2019 (COVID-19) and Need of Oxygen Support Without Mechanical Ventilation
Brief Title: Convalescent Antibodies Infusion in COVID 19 Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizative problems
Sponsor: Piero Luigi Ruggenenti (Other)
Collaborators: Aferetica (Unknown)
Responsible Party: Sponsor-Investigator, Piero Luigi Ruggenenti, Director, Unit of Nephrology, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFPP COVID 19 Early
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Pneumonia, Viral; Corona Virus Infection
Keywords: Pneumonia viral; COVID 19; Double-filtration plasmapheresis; Convalescent antibodies
MeSH Terms: conditions — Pneumonia, Viral; Coronavirus Infections; COVID-19 | interventions — Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental antibodies (immunoglobulins) infusion (Experimental): Anti-coronavirus obtained with double-filtration plasmapheresis (DFPP) from convalescent patients
  Interventions: Biological: Anti-coronavirus antibodies (immunoglobulins) obtained with DFPP form convalescent patients

INTERVENTIONS:
Biological: Anti-coronavirus antibodies (immunoglobulins) obtained with DFPP form convalescent patients — Antibodies obtained from consenting convalescent donors will be administered to ten consecutive patients who fulfill the inclusion criteria .

SUMMARY:
The outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which originated in Wuhan, China, has become a major concern all over the world.

Convalescent plasma or immunoglobulins have been used as a last resort to improve the survival rate of patients with SARS whose condition continued to deteriorate despite treatment with pulsed methylprednisolone. Moreover, several studies showed a shorter hospital stay and lower mortality in patients treated with convalescent plasma than those who were not treated with convalescent plasma. Evidence shows that convalescent plasma from patients who have recovered from viral infections can be used effectively as a treatment of patients with active disease.

The use of solutions enriched of antiviral antibodies has several important advantages over the convalescent plasma including the high level of neutralizing antibodies supplied. Moreover, plasma-exchange is expensive and requires large volumes of substitution fluid With either albumin or fresh frozen plasma, increasing the risk of cardiovascular instability in the plasma donor and in the recipient, which can be detrimental in a critically ill patient with COVID 19 pneumonia. The use of plasma as a substitution fluid further increases treatment costs and is associated with risk of infections, allergic reactions and citrate-induced hypocalcemia. Albumin is better tolerated and less expensive, but exchanges using albumin solutions increase the risk of bleeding because of progressive coagulation factor depletion.

The aforementioned limitations of plasma therapy can be in part overcome by using selective apheresis methods, such as double-filtration plasmapheresis (DFPP)3. During DFPP, plasma is separated from cellular components by a plasma filter, and is then allowed to pass through a fractionator filter. Depending on the membrane cut-off, the fractionator filter retains larger molecules and returns fluid along with smaller molecules to the circulation. Thus, the selection of a membrane with an appropriate sieving coefficient for IgG allows to efficiently clear autoantibodies in patients with antibody-mediated diseases (e.g., macroglobulinemia, myasthenia gravis and rheumatoid arthritis) with negligible fluid losses and limited removal of albumin and coagulation factors1.

In patients with severe membranous nephropathy and high titer of autoreactive, nephritogenic antibodies against the podocyte-expressed M type phospholipase A2 receptor (PLA2R), DFPP accelerated anti PLA2R depletion4. Measurement of the antibody titer in treated patient and recovered fluid showed that antibody removal was extremely effective and that large part of antibodies was removed during the first DFPP procedure. This therapeutic regimen was safe and well tolerated and easy to apply4. In an ongoing pilot study we found that the same methodological approach can be used to remove circulating antibodies from patients who recovered from COVID 19 and to infuse these antibodies in patients with active viral infection. Treatment was well tolerated and preliminary findings are encouraging. Thus, in this novel pilot study we aim to explore whether the infusion of antibodies obtained with one single DFPP procedure from voluntary convalescent donors could offer an effective and safe therapeutic option for patients with earlier stages of coronavirus (COVID-19) pneumonia requiring oxygen supply without mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

Plasma Ig Donors

* Adult (>18 and <65-yr-old) men and women
* Convalescent donor who recovered from COVID 19 from at least 14 days according to the clinical and laboratory criteria defined by the Consiglio Superiore di Sanità on February 20, 2019 ("The recovered patient is the one who resolves the symptoms of COVID-19 infection and who is negative in two consecutive tests for the search for SARS-Cov-2, performed 24 hours apart") with the exceptions mentioned in the attached derogation (that is "no upper age limit to donation provided there are no clinical contraindications to the procedure and independent of documented evidence of two negative tests for SARS-Cov 2 naso-faringeal contamination")
* Male or female donor; if female only if nulliparous; in both cases with a negative history of blood component transfusions
* Careful clinical evaluation of the patient-donor with particular reference to the criteria established by current legislation to protect the health of the donor who donates by apheresis
* Presence of adequate levels of neutralizing anti-SARS-COV-2 antibodies;
* Biological qualification test negative defined by current indications (performed at SIMT of HPG23)
* Test negative for: HAV RNA, HEV RNA, PVB19 DNA (performed at HPG23)
* Informed written consent

Recipients

* >18 years of age
* COVID-19 pneumonia diagnosed by standard criteria (viral detection in naso-faringeal or bronco-alveolar lavage by RT-PCR for SARS-COV-2, typical Chest X Ray or CT Scan, ventilatory dysfunction not directly explained by heart failure or fluid overload)
* Respiratory failure (i.e. room air PaO2<60 mmHg) needing oxygen support with Venturi mask (FiO2 between 28 and 60%), non-rebreathing mask or high flow-nasal cannula (HFNC);
* Patient written informed consent

Exclusion Criteria:

* Need of Continuous Positive Airway Pressure (CPAP) ventilator support, Non-Invasive Ventilation (NIV) or intubation for invasive mechanical ventilation
* Involvement in any clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Time to weaning of oxygen support | Through study completion, an average of 3 months

SECONDARY OUTCOMES:
Chest XR or CT scan evaluation | Changes during the study up completion, an average of 3 months
Survival, | Through study completion, an average of 3 months
Viral titer | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
Anti COVID 19 IgG antibodies | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
Anti COVID 19 IgM antibodies | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
C5a concentration | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
C3a concentration | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum C5b-9 concentration Marker of complement activation | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IL-6 levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IL-1b levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IFNγ levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum MCP-1 levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum TNFα levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IL-10 levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IL-2 levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.
Serum IL-7 levels | Changes from before Ig administration, one day after Ig administration and every week through study completion, an average of 3 months.
  Marker of complement activation in plasma.

IPD SHARING:
Plan to Share IPD: Undecided